CLINICAL TRIAL: NCT03594136
Title: Challenging Reference Values for Intracranial Pressure: A Prospective, Multicenter, Clinical Study
Brief Title: New Reference Values for Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Nicolas Alexander Norager, Researh Assistant, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P1NICP
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Intracranial Pressure
Keywords: Intracranial pressure; ICP; Normal value; Reference value; Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemetric intracranial pressure implant (Experimental): A telemetric intracranial pressure monitoring sensor is inserted into the brain parenchyma at the end of an uncomplicated surgery for an unruptured aneurysm
  Interventions: Device: Raumedic Neurovent-P-tel

INTERVENTIONS:
Device: Raumedic Neurovent-P-tel — Insertion of a Neurovent-P-tel in adults to study normal intracranial pressure

SUMMARY:
Intracranial pressure is a cornerstone in neurosurgical care used in a variety of diseases. However currently, doubts regarding normal intracranial pressure exist. Few studies have investigated normal intracranial pressure in truly normal adults. The aim of this study is to investigate intracranial pressure in adults who have normal intracranial pressure physiology.

In this prospective, multicenter, clinical study, the intracranial pressure of 10 adults requiring surgery for an unruptured aneurysm will be investigated. These patients are thought to be normal in terms of intracranial pressure physiology. At the end of their surgery for an aneurysm, a telemetric intracranial pressure monitoring sensor will be implanted. Afterward, intracranial pressure curves will be obtained non-invasively 1., 14., 30 and 90 days after implantation. The intracranial pressure will be investigated in 5 different positions (supine, lumbar, upright sitting, standing and walking). Furthermore, a 24-hour measurement will be performed in their home environment, thus investigating intracranial pressure under daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Requiring surgery for a "cold" (unruptured) aneurysm

Exclusion Criteria:

* Current or previous examination or treatment for hydrocephalus
* Current or previous examination or treatment for idiopathic intracranial hypertension
* Previous operation with insertion of cerebrospinal fluid shunt
* Previous trauma with intracranial hemorrhage
* Global cerebral edema
* Increased infection risks
* Surgical complications during the primary operation
* Unable to understand patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Normal Intracranial Pressure Values | Each participants will be monitored for three months
  To determine reference values for intracranial pressure in healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Marianne, D.M.Sc., Study Director — Rigshospitalet, Denmark
Locations (3):
- Military University Hospital Prague, Prague, Czechia
- Denmark (2):
  - Rigshospitalet, Copenhagen, Copenhagen E
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norager NH, Lilja-Cyron A, Riedel CS, Holst AV, Pedersen SH, Juhler M. Intracranial pressure following surgery of an unruptured intracranial aneurysm-a model for normal intracranial pressure in humans. Fluids Barriers CNS. 2024 May 21;21(1):44. doi: 10.1186/s12987-024-00549-1. PMID 38773608